CLINICAL TRIAL: NCT01303679
Title: Phase III Randomized Multicenter Trial Comparing Continued Maintenance Therapy With the Bevacizumab + Taxane Versus Bevacizumab + Substituting Exemestane in Patients With Metastatic Breast Cancer or Locally Advanced With Estrogen Receptor Positive and Having at Least a Stable Disease After 16 to 18 Weeks of Treatment With Bevacizumab + Taxane.
Brief Title: 1st Line Treatment of Bevacizumab-Taxane vs Bevacizumab-Exemestane in Metastatic Breast Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Not reveal any significant difference between the 2 treatment arms
Sponsor: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Arobase (GINECO-BR107)
Record Dates: First submitted 2011-02-23; First posted 2011-02-25 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: First Line Metastatic Breast Cancer
Keywords: First line metastatic breast cancer; Positive estrogen receptors; Negative HER2 receptors; At least stable disease after 4 months of paclitaxel-bevcizumab induction chemotheray
MeSH Terms: interventions — Paclitaxel; Bevacizumab; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- paclitaxel-bevacizumab (Active Comparator): Paclitaxel, 80mg/m² at d1, d8, d15 bevacizumab, 10 mg/kg at d1, d15
  Interventions: Drug: Paclitaxel; Drug: Bevacizumab
- exemestane-bevacizumab (Experimental): exemestane, 25 mg daily dose bevacizumab, 15mg/kg every 3 weeks
  Interventions: Drug: Bevacizumab; Drug: Exemestane

INTERVENTIONS:
Drug: Paclitaxel — IV, 80mg/m² at d1, d8, d15
  Arms: paclitaxel-bevacizumab
Drug: Bevacizumab — IV, 10 mg/kg at d1, d15 or IV, 15 mg/kg every 3 weeks
Drug: Exemestane — daily 25 mg (1 pill) oral intake
  Arms: exemestane-bevacizumab

SUMMARY:
In first-line metastatic breast cancer, the bevacizumab-taxane to progression or toxicity, is currently the standard treatment. In patients expressing hormone receptors, it was shown that hormone therapy administered in maintenance after induction chemotherapy, could have a benefit regarding the progression-free survival. The investigators make the hypothesis that there would be interest to discontinue treatment with taxane after 4 months, and to begin hormone therapy while continuing maintenance bevacizumab.

Exemestane was chosen because it has been shown potentially active in patients who progressed after letrozole, anastrozole or tamoxifen.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 ans.
* Metastatic breast cancer or locally advanced
* RE+, HER2-
* Patient receiving paclitaxel-bevacizumab first line chemotherapy

Exclusion Criteria:

* Previous treatment by exemestane (both in adjuvant or metastatic treatment).
* 1st line of chemotherapy different thaan paclitaxel-bevacizumab.
* Treatment by paclitaxel-bevacizumab > 18 weeks.
* HER2 positifs et/ou récepteurs aux oestrogènes négatifs.
* Previous thrombosis event within the 6 months before inclusion .
* Previous significant surgery within the 28 days before treatment start
* Previuous coagulopathy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2010-06; Primary Completion 2014-06 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Primary free survival | 24 months for recruitment and 18 months for follow up

CONTACTS AND LOCATIONS:
Overall Officials: Thomas BACHELOT, Md, Principal Investigator — GINECO
Locations (1):
- BACHELOT, Lyon, France

REFERENCES:
- [Derived] Tredan O, Follana P, Moullet I, Cropet C, Trager-Maury S, Dauba J, Lavau-Denes S, Dieras V, Beal-Ardisson D, Gouttebel M, Orfeuvre H, Stefani L, Jouannaud C, Burki F, Petit T, Guardiola E, Becuwe C, Blot E, Pujade-Lauraine E, Bachelot T. A phase III trial of exemestane plus bevacizumab maintenance therapy in patients with metastatic breast cancer after first-line taxane and bevacizumab: a GINECO group study. Ann Oncol. 2016 Jun;27(6):1020-1029. doi: 10.1093/annonc/mdw077. Epub 2016 Feb 24. PMID 26916095